CLINICAL TRIAL: NCT02527707
Title: A Phase 2, Open-Label Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamic Activity of a Titrating-Dose Lonafarnib/Ritonavir in Patients Chronically Infected With Hepatitis Delta Virus
Brief Title: Titrating-Dose of Lonafarnib in Combination With Ritonavir
Acronym: LOWR-4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eiger BioPharmaceuticals (Industry)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EIG-LNF-002
Expanded Access: NCT03895528 (Approved for marketing)
Record Dates: First submitted 2015-08-13; First posted 2015-08-19 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Chronic Delta Hepatitis
MeSH Terms: conditions — Hepatitis D, Chronic | interventions — lonafarnib; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lonafarnib/ritonavir (Experimental): Lonafarnib starting at 50 mg BID in combination with ritonavir 100 mg BID and escalating to lonafarnib 75 mg BID and then 100 mg BID as tolerated. The duration of the study for each patient is 6 months of treatment and 6 months follow-up.
  Interventions: Drug: lonafarnib; Drug: Ritonavir

INTERVENTIONS:
Drug: lonafarnib — antiviral farnesyltransferase inhibitor
  Other Names: EBP994; Sarasar
Drug: Ritonavir — Cytochromes P450 3A4 inhibitor used to boost lonafarnib
  Other Names: Norvir

SUMMARY:
A phase 2, open-label study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamic activity of titrating-dose lonafarnib/ritonavir in patients chronically infected with hepatitis delta virus (HDV)

DETAILED DESCRIPTION:
This is a Phase 2 study of 24 weeks of treatment with a dose-titration regimen of lonafarnib/ritonavir in up to 15 patients chronically infected with HDV: lonafarnib starting at 50 mg twice daily (BID) in combination with ritonavir 100 mg BID and escalating lonafarnib as tolerated.

The duration of the study for each patient is approximately 13 months (up to 4 weeks for screening, 24 weeks of treatment, 4 weeks for the primary follow-up visit, and monthly safety follow-up visits for 5 months thereafter). The 6-month follow-up after the last dose of study drug is designed to allow evaluation of the clinical and virologic course after completion of the 24-week Treatment Period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, 18 to 65 years of age, inclusive
2. Chronic HDV infection documented by a positive HDV antibody (Ab) test of at least 6 months duration and detectable HDV ribonucleic acid (RNA) by quantitative polymerase chain reaction (qPCR) at study entry
3. Liver biopsy demonstrating evidence of chronic hepatitis
4. Willingness to practice appropriate contraception

Key Exclusion Criteria:

1. Previous use of lonafarnib
2. Co-infected with human immunodeficiency virus (HIV) or hepatitis C virus (HCV)
3. Active jaundice defined by total bilirubin level >2.0 mg/dL and known not to have Gilbert's disease
4. Decompensated liver disease or cirrhosis, history of bleeding esophageal varices, ascites, or hepatic encephalopathy
5. Serum creatinine concentration ≥1.5 times upper limit of normal (ULN)
6. Evidence of another form of viral hepatitis (not including hepatitis B virus or HCV) or another form of liver disease
7. Evidence of hepatocellular carcinoma
8. Use of alfa interferon, either interferon alfa-2a or interferon alfa-2b, or peginterferon alfa-2a within 2 months before the start of screening
9. Concomitant use of any of the following:

   1. Medications or foods that are known moderate or strong inducers or inhibitors of CYP3A4 or CYP2C19
   2. Drugs known to prolong the PR interval or QT interval of the electrocardiogram
   3. Receipt of systemic immunosuppressive therapy within the 3 months before start of screening
   4. Statins, due to inhibition of mevalonate synthesis, which reduces protein prenylation
   5. Medications contraindicated in the prescribing information for ritonavir

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2017-02-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heiner Wedemeyer, MD, PhD, Principal Investigator — Hannover Medical School

REFERENCES:
- [Background] Koh C, Canini L, Dahari H, Zhao X, Uprichard SL, Haynes-Williams V, Winters MA, Subramanya G, Cooper SL, Pinto P, Wolff EF, Bishop R, Ai Thanda Han M, Cotler SJ, Kleiner DE, Keskin O, Idilman R, Yurdaydin C, Glenn JS, Heller T. Oral prenylation inhibition with lonafarnib in chronic hepatitis D infection: a proof-of-concept randomised, double-blind, placebo-controlled phase 2A trial. Lancet Infect Dis. 2015 Oct;15(10):1167-1174. doi: 10.1016/S1473-3099(15)00074-2. Epub 2015 Jul 16. PMID 26189433
- [Background] Yurdaydin C, Keskin O, Kalkan C, Karakaya F, Caliskan A, Karatayli E, Karatayli S, Bozdayi AM, Koh C, Heller T, Idilman R, Glenn JS. Optimizing lonafarnib treatment for the management of chronic delta hepatitis: The LOWR HDV-1 study. Hepatology. 2018 Apr;67(4):1224-1236. doi: 10.1002/hep.29658. Epub 2018 Feb 19. PMID 29152762
- [Background] Yurdaydin C, Keskin O, Yurdcu E, Caliskan A, Onem S, Karakaya F, Kalkan C, Karatayli E, Karatayli S, Choong I, Apelian D, Koh C, Heller T, Idilman R, Bozdayi AM, Glenn JS. A phase 2 dose-finding study of lonafarnib and ritonavir with or without interferon alpha for chronic delta hepatitis. Hepatology. 2022 Jun;75(6):1551-1565. doi: 10.1002/hep.32259. Epub 2021 Dec 23. PMID 34860418
- See also: Eiger BioPharmaceuticals, Inc. company website — http://eigerbio.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Lonafarnib/Ritonavir: Lonafarnib starting at 50 mg twice daily (BID) in combination with ritonavir 100 mg BID and escalating to lonafarnib 75 mg BID and then 100 mg BID as tolerated. The duration of the study for each patient is 6 months of treatment and 6 months follow-up.
  lonafarnib: antiviral farnesyltransferase inhibitor
  Ritonavir: Cytochromes P450 3A4 inhibitor used to boost lonafarnib
Period: Overall Study
Arm/Group | Lonafarnib/Ritonavir
Started | 15
Completed | 13
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Lonafarnib/Ritonavir
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 42 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 in Mean Hepatitis D Virus (HDV) Ribonucleic Acid (RNA) Titer
Description: Change from baseline to Week 24 in mean HDV RNA titer following dose escalating from lonafarnib 50 mg BID to 75 mg BID and to 100 mg BID, all boosted with ritonavir 100 mg BID.
Time Frame: Baseline and Week 24 (6 months)
Measure: Mean (Standard Deviation); unit: log IU/mL
Arm/Group | Lonafarnib/Ritonavir
Number analyzed (Participants) | 15
log IU/mL | -1.62 (1.4)

2. Secondary Outcome: Number of Patients With 1 Log Reduction From Baseline by Timepoint
Description: Number of patients with at least 1 log reduction in HDV RNA from baseline by dose level and timepoint
Time Frame: Baseline and Week 1, Week 2, Week 4, Week 6, Week 8, Week 12, Week 16, Week 20, or Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Lonafarnib/Ritonavir
Number analyzed (Participants) | 13
Participants
  Week 1 | 7
  Week 2 | 6
  Week 4 | 10
  Week 6 | 11
  Week 8 | 10
  Week 12 | 12
  Week 16 | 12
  Week 20 | 10
  Week 24 | 9

ADVERSE EVENTS:
Time Frame: 6 months on treatment, 6 months off-treatment follow-up.
Arm/Group | Lonafarnib/Ritonavir
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonafarnib/Ritonavir (N=15)
mandibular fracture) (Injury, poisoning and procedural complications) | 1 (1) — Patient involved in a fight where he sustained a mandibular fracture and was hospitalized. The investigator considered the event not to be related to lonafarnib or ritonavir.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lonafarnib/Ritonavir (N=15)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 15 (15)
Nausea (Gastrointestinal disorders) | 8 (8)
Vomiting (Gastrointestinal disorders) | 8 (8)
Abdominal Pain (Gastrointestinal disorders) | 6 (6)
Fatigue (General disorders) | 4 (4)
Asthenia (General disorders) | 3 (3)
Weight Decrease (Investigations) | 8 (8)
Decrease Appetite (Metabolism and nutrition disorders) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 4 (4)
Dizziness (Nervous system disorders) | 4 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Acne (Skin and subcutaneous tissue disorders) | 2 (2)
Pruitis (Skin and subcutaneous tissue disorders) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 2 (2)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-22): https://cdn.clinicaltrials.gov/large-docs/07/NCT02527707/Prot_000.pdf
  • Statistical Analysis Plan (2016-09-21): https://cdn.clinicaltrials.gov/large-docs/07/NCT02527707/SAP_001.pdf